CLINICAL TRIAL: NCT07052942
Title: Individualizing Treatment for Asthma in Primary Care (Full Study)
Acronym: iTREAT-PC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: DARTNet Institute (Other Government)
Collaborators: Penn State University (Other); Icahn School of Medicine at Mount Sinai (Other); University of Colorado, Denver (Other); RAND (Other); University of Washington (Other); University of North Carolina (Other); Reliant Medical Group (Other); Kelsey Research Foundation (Other); University of Kansas (Other); University of Missouri-Columbia (Other); John Peter Smith Health Network (Unknown); Rutgers University (Other); AdventHealth (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLACER-2021C3-24737-IC_Full; PLACER-2021C3-24737-IC_Full (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Asthma; Asthma Attack; Asthma Exacerbations
Keywords: Intervention/Treatment
MeSH Terms: conditions — Asthma | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: The investigators are intentionally avoiding the factorial design framework for the purpose of analysis. This is because the investigators are uncertain about whether the combined treatments will have an additive effect. If the combined effect is less than additive, then the standard main effects analysis based on the factorial design is not optimal. The primary analysis will consist of three hypothesis tests comparing each of the three treatment arms against the control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Inhaled corticosteroids as part of rescue therapy (R-ICS) (Active Comparator): Maintenance And Reliever Therapy (MART), or Patient Activated Reliever Triggered Inhaled Corticosteroids (PARTICS) - this includes budesonide-albuterol (AirSupra)
  Interventions: Drug: Inhaled corticosteroid (ICS); Other: Asthma Symptom Monitoring Web-based Application
- Azithromycin (AZ) (Active Comparator): Azithromycin - 500mg three times per week. Can be reduced to 250 mg three times per week for side effects.
  Interventions: Drug: Azithromycin; Other: Asthma Symptom Monitoring Web-based Application
- Enhanced Usual Care (Other): Participants will be asked to use an online Asthma Symptom Monitoring (ASM) tool to enhance communication with the medical team as well as self-awareness of their asthma symptoms. There are no "study drugs" in this intervention.
  Interventions: Other: Asthma Symptom Monitoring Web-based Application
- Inhaled corticosteroids as part of rescue therapy (R-ICS) + Azithromycin (Active Comparator): R-ICS either as MART therapy or PARTICS + Azithromycin
  Interventions: Drug: Inhaled corticosteroid (ICS); Drug: Azithromycin; Other: Asthma Symptom Monitoring Web-based Application

INTERVENTIONS:
Drug: Inhaled corticosteroid (ICS) — Participants will use either a combination of budesonide/formoterol or mometasone/formoterol as both controller and rescue therapy or a stand alone inhaled steroid (beclomethasone, budesonide, fluticasone, mometasone, ciclesodine) of their choice with their current reliever therapy or be converted to budesonide/albuterol as rescue therapy.
  Arms: Inhaled corticosteroids as part of rescue therapy (R-ICS); Inhaled corticosteroids as part of rescue therapy (R-ICS) + Azithromycin
Drug: Azithromycin — Participants will take 500mg of azithromycin three times a week or 10mg/kg if under 50Kg which may be reduced to 250mg/Kg for side effects.
  Arms: Azithromycin (AZ); Inhaled corticosteroids as part of rescue therapy (R-ICS) + Azithromycin
Other: Asthma Symptom Monitoring Web-based Application — All participants will be provided access to the Asthma Symptom Monitoring (ASM) tools. ASM can be integrated with electronic health records (EHR) or used as a stand alone application. Participants will answer 5 questions about their asthma each week. If symptoms are problematic, participants can request a call back from a person on their care team. Participants can view a graph of their data, watch videos, and record peak flows. Clinicians and members of the care team can view data in the EHR (not for stand alone web app).

SUMMARY:
While asthma therapy is becoming more individualized based on asthma phenotypes, more research is needed to tailor newer therapies to individuals. Inhaled corticosteroid (ICS) medications are the foundation of care for all individuals with persistent asthma. But ICS use is not without possible long term side effects.

This study will compare two currently available approaches to reduce AEX in primary care patients: (1) use of inhaled corticosteroids (ICS) as part of rescue therapy, also known as MART (Maintenance And Reliever Therapy) or PARTICS (Patient Activated Reliever Trigger Inhaled Corticosteriods) therapy - either of these therapies will be called Rescue-Inhaled Corticosteroids or R-ICS pronounced "Ricks," and (2) use of azithromycin (AZ) as a preventive therapy. These treatments will be studied both individually and in combination.

DETAILED DESCRIPTION:
Design. Four arm, patient level randomized trial (N=3200). Comparators: Rescue inhaled corticosteroids (R-ICS) versus azithromycin versus R-ICS plus azithromycin versus control patients. All arms will include home monitoring of asthma symptoms using various web application approaches. R-ICS therapy will consist of a corticosteriod/formoterol inhaler, a stand-alone ICS inhaler used with usual rescue therapy or when available a combination corticosteroid/albuterol inhaler, the initial azithromycin dose will be 500mg (10mg/Kg) three times a week and may be titrated down to 250mg (10mg/Kg) three times per week for side effects. Exacerbations will be blindly adjudicated. Individuals who experience three exacerbations in < 12 months will have their treatments "stepped-up,"unless in the dual treatment arm; control participants going to R-ICS and single therapy participants to dual therapy. Individuals completing either of the azithromycin arms will be offered up to 12 additional months of follow-up after stopping the azithromycin only.

ELIGIBILITY:
Inclusion Criteria:

1. A clinical asthma diagnosis for at least 1 year;
2. 13-75 years of age;
3. A prescription for an ICS either used regularly, or on an as needed controller, not reliever, schedule - ICS or ICS + LABA or ICS+LABA+LAMA;
4. A current ACT total score of <20 OR an exacerbation requiring 72 hours or more of systemic steroids or a hospitalization of at least 24 hours > 30 days and < 365 days prior to enrollment;
5. Able to provide consent (adolescents: assent) in English or Spanish; (i.e., cognitively impaired individuals are deemed not to be able to provide consent and thus do not meet inclusion criteria.);
6. Patients with a coexisting clinical diagnosis of COPD are eligible if they meet any one of the following criteria:

   (i) Never smoker without secondary lung disease causing airway obstruction. (ii) Current or former smoker with obstruction on PFTs, but normal diffusing capacity of the lungs for carbon monoxide (DLCO) in the past 24 months.
7. Patients on medications that may interact with azithromycin but are not totally excluded may be enrolled if they agree to a cardiac rhythm strip after consent and prior to randomization (or have an ECG within the prior 24 months as a baseline assessment) and a repeat rhythm strip after one week if randomized to one of the azithromycin arms of the study.

Exclusion Criteria:

1. Another family member living in the same household already enrolled in study;
2. Life expectancy <1 year (operationalized by the question to the patient's asthma care clinician "Would you be surprised if this person died in the next 12 months? If yes - include, if no - exclude);
3. No ICS prescribed for the individual (does not have to be using the ICS inhaler);
4. Active treatment for hematological or solid organ cancer other than basal cell or skin squamous cell cancer (if participant is > 12 months out from original therapy and may be on a cancer maintenance drug that is not otherwise contraindicated they are eligible for the study);
5. Allergy to macrolides or conditions for which macrolide administration may possibly be hazardous (e.g., acute or chronic hepatitis, cirrhosis, or other liver disease; end-stage renal disease; uncorrected hypokalemia or hypomagnesemia; clinically significant bradycardia; or history of prolonged cardiac repolarization and QT interval or evidence of prolonged cardiac repolarization on rhythm strip and QT interval or torsades de pointes);
6. On daily or every other day oral steroids for any reason;
7. A course of systemic steroids for an asthma exacerbation or an overnight hospitalization for an asthma exacerbation in the past month (can wait and re-check eligibility after one month);
8. Currently on R-ICS or any antibiotic therapy expected to last more than 30 days. If on antibiotics less than 30 days, individual can enroll after they have stopped their current antibiotic for 72 hours. Individuals on biologics can be enrolled if they have been on a stable dose for > 6 months and meet the ACT or exacerbation criteria as well as all other criteria after being on the stable does of the biologic.
9. On a medication with known risk (i.e., that is associated with prolonged QT and associated with torsades de pointes even when taken as recommended)- absolute contraindication to eligibility- Full lists in Appendix B;
10. Specified medications for which close monitoring has been recommended in the setting of macrolide administration (digoxin, warfarin, theophylline, ergotamine or dihydroergotamine, cyclosporine, hexobarbital, phenytoin or nelfinavir).

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2029-11-15 (Estimated); Study Completion 2029-11-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Asthma Exacerbations Per Year | Follow-up is up to 16 months.
  The primary outcome, the rate of asthma exacerbations per year, is defined as the number of exacerbations, emergency room visits, or hospitalizations requiring oral or parenteral corticosteroids, per patient per year, monthly through study completion.

SECONDARY OUTCOMES:
Asthma Control as Measured by the Asthma Control Test (ACT) | Follow-up is up to 16 months.
  Asthma control represents the degree to which impairment (impact of asthma on patient's daily life) is minimized and the goals of therapy are met. The Asthma Control Test is a participant administered tool for assessing the level of asthma control. Total scores range from 5 to 25, with a score of 20 to 25 indicating well-controlled asthma, a score of 16 to 19 indicating asthma that was not well controlled, and a score of 5 to 15 indicating very poorly controlled asthma. The Asthma Control Test has a score range of 5 to 25 with higher scores indicating better control.
Asthma Quality of Life Questionnaire (AQLQ) as Measured by the Juniper Mini Asthma Quality of Life Questionnaire | Follow-up is up to 16 months.
  The Asthma Quality of Life Questionnaire is a participant-administered tool for assessing functional impairment. Total scores range from 1 to 7, with a score of 7=no impairment and 1=maximum impairment.
Days Per Year Lost From Work or School/ Days Unable to Carry Out Usual Activities Due to Asthma | Follow-up is up to 16 months.
  Defined as days not able to work or go to school because of asthma symptoms OR days not able to carry out usual activities due to asthma.

CONTACTS AND LOCATIONS:
Overall Officials: Wilson D Pace, MD, FAAFP, Principal Investigator — DARTNet Institute; Dave Mauger, PhD, Principal Investigator — Penn State University
Locations (13):
- United States (13):
  - DARTNet Institute, Aurora, Colorado
  - University Colorado-Denver, Aurora, Colorado
  - AdventHealth, Orlando, Florida
  - University of Kansas, Kansas City, Kansas
  - Reliant Medical Group, Worcester, Massachusetts
  - University of Missouri, Columbia, Missouri
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Mt. Sinai School of Medicine, New York, New York
  - University North Carolina, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - JPS Health Network, Fort Worth, Texas
  - Kelsey Research Foundation, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Analyzable data set will be submitted to PCORI at the conclusion of the study. This will include the final cleaned and locked data set that contains all the data used in conducting the analyses reported in the PCORI Final Research Report and is de-identified in accordance with the HIPAA Privacy. Rule (45 C.F.R. § 164.514(b)).
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Anticipated date is no later than 6/31/31.
Access Criteria: Users interested in obtaining study data will need to complete a Restricted Data Use Agreement, specify the reason for the request, and obtain IRB approval or notice of exemption for their research.
URL: https://www.pcori.org/about/governance/pcoris-policy-data-management-and-data-sharing

REFERENCES:
- [Background] Global Initiative for Asthma. Global strategy for asthma management and prevention 2023 report. Accessed February 10, 2024. https://ginasthma.org/2023-gina-main-report/
- [Background] Calmes D, Huynen P, Paulus V, Henket M, Guissard F, Moermans C, Louis R, Schleich F. Chronic infection with Chlamydia pneumoniae in asthma: a type-2 low infection related phenotype. Respir Res. 2021 Feb 26;22(1):72. doi: 10.1186/s12931-021-01635-w. PMID 33637072
- [Background] Wenzel SE. Severe Adult Asthmas: Integrating Clinical Features, Biology, and Therapeutics to Improve Outcomes. Am J Respir Crit Care Med. 2021 Apr 1;203(7):809-821. doi: 10.1164/rccm.202009-3631CI. PMID 33326352
- [Background] Ray A, Camiolo M, Fitzpatrick A, Gauthier M, Wenzel SE. Are We Meeting the Promise of Endotypes and Precision Medicine in Asthma? Physiol Rev. 2020 Jul 1;100(3):983-1017. doi: 10.1152/physrev.00023.2019. Epub 2020 Jan 9. PMID 31917651
- [Background] Israel E, Cardet JC, Carroll JK, Fuhlbrigge AL, She L, Rockhold FW, Maher NE, Fagan M, Forth VE, Yawn BP, Arias Hernandez P, Kruse JM, Manning BK, Rodriguez-Louis J, Shields JB, Ericson B, Colon-Moya AD, Madison S, Coyne-Beasley T, Hammer GM, Kaplan BM, Rand CS, Robles J, Thompson O, Wechsler ME, Wisnivesky JP, McKee MD, Jariwala SP, Jerschow E, Busse PJ, Kaelber DC, Nazario S, Hernandez ML, Apter AJ, Chang KL, Pinto-Plata V, Stranges PM, Hurley LP, Trevor J, Casale TB, Chupp G, Riley IL, Shenoy K, Pasarica M, Calderon-Candelario RA, Tapp H, Baydur A, Pace WD. Reliever-Triggered Inhaled Glucocorticoid in Black and Latinx Adults with Asthma. N Engl J Med. 2022 Apr 21;386(16):1505-1518. doi: 10.1056/NEJMoa2118813. Epub 2022 Feb 26. PMID 35213105